CLINICAL TRIAL: NCT05433701
Title: A Phase III Randomized Controlled Non-inferiority Trial to Compare Stereotactic Body Radiotherapy Versus Radiofrequency Ablation for Unresectable, Small (≤ 3 cm) Hepatocellular Carcinoma
Brief Title: Stereotactic Body Radiotherapy Versus Radiofrequency Ablation for Unresectable, Small (≤ 3 cm) HCC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonggi Choi (Other)
Responsible Party: Sponsor-Investigator, Jonggi Choi, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STR_1
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFA group (Active Comparator): * RFA are performed under local anesthesia or monitored anesthesia care with either a 15-gause or 17-gause internally cooled electrode, depending on the size of the tumor.
  * RFA procedures are continued by modifying the output power based on the location and size of the tumor until the entire tumor and border area sizes of greater than 0.5 cm are included in the detected target lesion on ultrasound or CT.
  Interventions: Procedure: Radiofrequency Ablation
- SBRT group (Experimental): A total dose of 45 Gy is presecribed using 15 Gy per fraction over 3 consecutive days.
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — * Verify the setup position and respiration of patients as in the simulation CT image.
  * To precisely align the tumor prior to each treatment, cone-beam CT and gated fluoroscopy using the On-board Imager mounted on the linear accelerator are performed.
  * The Real-time Position Management system is used to monitor the accuracy of breathing phase during treatment.
  Arms: SBRT group
Procedure: Radiofrequency Ablation — - RFA are performed under local anesthesia or monitored anesthesia care with either a 15-gause or 17-gause internally cooled electrode, depending on the size of the tumor.
  Arms: RFA group

SUMMARY:
Hepatocellular carcinoma (HCC) is the third leading cause of cancer-related mortality and the sixth most prevalent cancer in the world. Standard treatments for early-stage HCCs include resection, liver transplantation, and percutaneous ablation, with 5-year survival rates of over 50 percent. Less than one-third of patients, however, are candidates for hepatic resection, and the use of radiofrequency ablation (RFA) may be significantly limited in cases with unfavorable tumor location and poor visibility on images, which increase the risk of technical failures and complications after RFA.

Recent advancements in radiotherapy and imaging have made it possible to deliver optimal radiation doses on the tumor site while minimizing exposure to normal organs. Stereotactic body radiation therapy (SBRT) is a method of high-precision radiation therapy that concentrates high-dose radiation to HCC in a short period of time to maximize the therapeutic effect on the tumor and minimize the side effects on normal tissues. Prospective and retrospective studies on SBRT for HCC have demonstrated its efficacy for local tumor control in small HCC. On the basis of these promising clinical results, a number of studies have compared the efficacy of RFA and SBRT. However, there is no strong evidence from randomized controlled trials comparing SBRT and RFA.

In order to evaluate and compare the local efficacy and clinical outcomes of SBRT and RFA in patients with recurrent HCC, we conduct this non-inferiority trial.

DETAILED DESCRIPTION:
A total of 178 subjects are randomly assigned to one of two treatment groups (89 patients in the body stereotactic radiotherapy group and 89 patients in the radiofrequency ablation group). If the assigned treatment method is technically infeasible, patients are allowed to be treated with the other method.

* RFA: When localization of the lesion is difficult under image guidance, when it is difficult to secure a safe needle path, when there is a risk of collateral thermal damage to adjacent organs, and when it is difficult to prevent it.
* SBRT: When irradiation with 45 Gy (daily dose of 15 Gy) is infeasible due to the maximum tolerance dose of normal organs.

ELIGIBILITY:
Inclusion Criteria:

1. patient over the age of 18
2. primary or recurrent HCC that is not suitable for surgery
3. HCCs with a longest diameter of ≤3cm and ≤2 lesions
4. no evidence of intrahepatic or extrahepatic residual disease except for target lesions
5. Child-Pugh class A or B hepatic function
6. no macroscopic vascular invasion or extrahepatic metastasis
7. written informed consent

Exclusion Criteria:

1. Eastern Cooperative Oncology Group performance status score 3 or 4
2. uncontrolled ascites, variceal bleeding, or hepatic encephalopathy
3. previous history of liver transplantation
4. an active gastric or duodenal ulcer within 3 months before screening
5. pregnant woman
6. uncontrolled other malignancies except for HCC within 2 years before screening
7. platelet count <50,000/µl
8. Patients who are judged by the researcher to be difficult to conduct clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Local progression-free survival rate, per-protocol (PP) | At year 2
  Local progression-free survival rate, PP

SECONDARY OUTCOMES:
Progression-free survival rate, intention-to-treat (ITT) | At year 2
  Progression-free survival rate, intention-to-treat (ITT)
Overall survival rate, ITT | At year 2
  Overall survival rate, ITT
Intrahepatic progression-free survival rate, PP | At year 2
  Intrahepatic progression-free survival rate, PP
Intrahepatic progression-free survival rate, ITT | At year 2
  Intrahepatic progression-free survival rate, ITT
Progression-free survival rate, PP | At year 2
  Progression-free survival rate, PP
Progression-free survival rate, ITT | At year 2
  progression-free survival rate, ITT
Adverse reaction rate, PP | At year 2
  Adverse reaction rate, PP
Adverse reaction rate, ITT | At year 2
  adverse reaction rate, ITT
Adverse reaction rate ≥ Gr 3, PP | At year 2
  Adverse reaction rate ≥ Gr 3, PP
Adverse reaction rate ≥ Gr 3, ITT | At year 2
  Adverse reaction rate ≥ Gr 3, ITT
Change of Child-Pugh score , PP | At year 2
  Change of Child-Pugh score , PP
Change of Child-Pugh score, ITT | At year 2
  Change of Child-Pugh score, ITT
Local progression-free survival rate according to the tumor location, PP | At year 2
  Local progression-free survival rate according to the tumor location, PP
Local progression-free survival rate according to the tumor location, ITT | At year 2
  Local progression-free survival rate according to the tumor location, ITT

CONTACTS AND LOCATIONS:
Overall Officials: Jonggi Choi, M.D, Ph D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erratum: Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2020 Jul;70(4):313. doi: 10.3322/caac.21609. Epub 2020 Apr 6. No abstract available. PMID 32767693
- [Background] Reig M, Forner A, Rimola J, Ferrer-Fabrega J, Burrel M, Garcia-Criado A, Kelley RK, Galle PR, Mazzaferro V, Salem R, Sangro B, Singal AG, Vogel A, Fuster J, Ayuso C, Bruix J. BCLC strategy for prognosis prediction and treatment recommendation: The 2022 update. J Hepatol. 2022 Mar;76(3):681-693. doi: 10.1016/j.jhep.2021.11.018. Epub 2021 Nov 19. PMID 34801630
- [Background] Lau WY, Lai EC. Salvage surgery following downstaging of unresectable hepatocellular carcinoma--a strategy to increase resectability. Ann Surg Oncol. 2007 Dec;14(12):3301-9. doi: 10.1245/s10434-007-9549-7. Epub 2007 Sep 22. PMID 17891443
- [Background] Chen MS, Li JQ, Zheng Y, Guo RP, Liang HH, Zhang YQ, Lin XJ, Lau WY. A prospective randomized trial comparing percutaneous local ablative therapy and partial hepatectomy for small hepatocellular carcinoma. Ann Surg. 2006 Mar;243(3):321-8. doi: 10.1097/01.sla.0000201480.65519.b8. PMID 16495695
- [Background] Feng K, Yan J, Li X, Xia F, Ma K, Wang S, Bie P, Dong J. A randomized controlled trial of radiofrequency ablation and surgical resection in the treatment of small hepatocellular carcinoma. J Hepatol. 2012 Oct;57(4):794-802. doi: 10.1016/j.jhep.2012.05.007. Epub 2012 May 23. PMID 22634125
- [Background] Huang J, Yan L, Cheng Z, Wu H, Du L, Wang J, Xu Y, Zeng Y. A randomized trial comparing radiofrequency ablation and surgical resection for HCC conforming to the Milan criteria. Ann Surg. 2010 Dec;252(6):903-12. doi: 10.1097/SLA.0b013e3181efc656. PMID 21107100
- [Background] Liu PH, Hsu CY, Hsia CY, Lee YH, Huang YH, Chiou YY, Lin HC, Huo TI. Surgical Resection Versus Radiofrequency Ablation for Single Hepatocellular Carcinoma </= 2 cm in a Propensity Score Model. Ann Surg. 2016 Mar;263(3):538-45. doi: 10.1097/SLA.0000000000001178. PMID 25775062
- [Background] Taguchi H, Sakuhara Y, Hige S, Kitamura K, Osaka Y, Abo D, Uchida D, Sawada A, Kamiyama T, Shimizu T, Shirato H, Miyasaka K. Intercepting radiotherapy using a real-time tumor-tracking radiotherapy system for highly selected patients with hepatocellular carcinoma unresectable with other modalities. Int J Radiat Oncol Biol Phys. 2007 Oct 1;69(2):376-80. doi: 10.1016/j.ijrobp.2007.03.042. PMID 17869660
- [Background] Krishnan S, Dawson LA, Seong J, Akine Y, Beddar S, Briere TM, Crane CH, Mornex F. Radiotherapy for hepatocellular carcinoma: an overview. Ann Surg Oncol. 2008 Apr;15(4):1015-24. doi: 10.1245/s10434-007-9729-5. Epub 2008 Jan 31. No abstract available. PMID 18236114
- [Background] Tse RV, Guha C, Dawson LA. Conformal radiotherapy for hepatocellular carcinoma. Crit Rev Oncol Hematol. 2008 Aug;67(2):113-23. doi: 10.1016/j.critrevonc.2008.01.005. Epub 2008 Mar 4. PMID 18308583
- [Background] Jeong Y, Jung J, Cho B, Kwak J, Jeong C, Kim JH, Park JH, Kim SY, Shim JH, Kim KM, Lim YS, Lee HC, Yoon SM. Stereotactic body radiation therapy using a respiratory-gated volumetric-modulated arc therapy technique for small hepatocellular carcinoma. BMC Cancer. 2018 Apr 13;18(1):416. doi: 10.1186/s12885-018-4340-7. PMID 29653562
- [Background] Takeda A, Sanuki N, Tsurugai Y, Iwabuchi S, Matsunaga K, Ebinuma H, Imajo K, Aoki Y, Saito H, Kunieda E. Phase 2 study of stereotactic body radiotherapy and optional transarterial chemoembolization for solitary hepatocellular carcinoma not amenable to resection and radiofrequency ablation. Cancer. 2016 Jul 1;122(13):2041-9. doi: 10.1002/cncr.30008. Epub 2016 Apr 8. PMID 27062278
- [Background] Su TS, Liang P, Lu HZ, Liang J, Gao YC, Zhou Y, Huang Y, Tang MY, Liang JN. Stereotactic body radiation therapy for small primary or recurrent hepatocellular carcinoma in 132 Chinese patients. J Surg Oncol. 2016 Feb;113(2):181-7. doi: 10.1002/jso.24128. Epub 2015 Dec 14. PMID 26799260
- [Background] Kimura T, Aikata H, Takahashi S, Takahashi I, Nishibuchi I, Doi Y, Kenjo M, Murakami Y, Honda Y, Kakizawa H, Awai K, Chayama K, Nagata Y. Stereotactic body radiotherapy for patients with small hepatocellular carcinoma ineligible for resection or ablation therapies. Hepatol Res. 2015 Apr;45(4):378-86. doi: 10.1111/hepr.12359. Epub 2014 Jun 16. PMID 24849379
- [Background] Takeda A, Sanuki N, Eriguchi T, Kobayashi T, Iwabutchi S, Matsunaga K, Mizuno T, Yashiro K, Nisimura S, Kunieda E. Stereotactic ablative body radiotherapy for previously untreated solitary hepatocellular carcinoma. J Gastroenterol Hepatol. 2014 Feb;29(2):372-9. doi: 10.1111/jgh.12350. PMID 23927053
- [Background] Jung J, Yoon SM, Kim SY, Cho B, Park JH, Kim SS, Song SY, Lee SW, Ahn SD, Choi EK, Kim JH. Radiation-induced liver disease after stereotactic body radiotherapy for small hepatocellular carcinoma: clinical and dose-volumetric parameters. Radiat Oncol. 2013 Oct 27;8:249. doi: 10.1186/1748-717X-8-249. PMID 24160910
- [Background] Andolino DL, Johnson CS, Maluccio M, Kwo P, Tector AJ, Zook J, Johnstone PA, Cardenes HR. Stereotactic body radiotherapy for primary hepatocellular carcinoma. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e447-53. doi: 10.1016/j.ijrobp.2011.04.011. Epub 2011 Jun 7. PMID 21645977
- [Background] Wahl DR, Stenmark MH, Tao Y, Pollom EL, Caoili EM, Lawrence TS, Schipper MJ, Feng M. Outcomes After Stereotactic Body Radiotherapy or Radiofrequency Ablation for Hepatocellular Carcinoma. J Clin Oncol. 2016 Feb 10;34(5):452-9. doi: 10.1200/JCO.2015.61.4925. Epub 2015 Nov 30. PMID 26628466
- [Background] Kim TH, Koh YH, Kim BH, Kim MJ, Lee JH, Park B, Park JW. Proton beam radiotherapy vs. radiofrequency ablation for recurrent hepatocellular carcinoma: A randomized phase III trial. J Hepatol. 2021 Mar;74(3):603-612. doi: 10.1016/j.jhep.2020.09.026. Epub 2020 Oct 5. PMID 33031846
- [Background] Marrero JA, Kulik LM, Sirlin CB, Zhu AX, Finn RS, Abecassis MM, Roberts LR, Heimbach JK. Diagnosis, Staging, and Management of Hepatocellular Carcinoma: 2018 Practice Guidance by the American Association for the Study of Liver Diseases. Hepatology. 2018 Aug;68(2):723-750. doi: 10.1002/hep.29913. No abstract available. PMID 29624699
- [Background] Rhim H, Yoon KH, Lee JM, Cho Y, Cho JS, Kim SH, Lee WJ, Lim HK, Nam GJ, Han SS, Kim YH, Park CM, Kim PN, Byun JY. Major complications after radio-frequency thermal ablation of hepatic tumors: spectrum of imaging findings. Radiographics. 2003 Jan-Feb;23(1):123-34; discussion 134-6. doi: 10.1148/rg.231025054. PMID 12533647
- [Background] Takaki H, Yamakado K, Nakatsuka A, Yamada T, Shiraki K, Takei Y, Takeda K. Frequency of and risk factors for complications after liver radiofrequency ablation under CT fluoroscopic guidance in 1500 sessions: single-center experience. AJR Am J Roentgenol. 2013 Mar;200(3):658-64. doi: 10.2214/AJR.12.8691. PMID 23436859